CLINICAL TRIAL: NCT02050958
Title: A Randomised, Open Label, Evaluator Blinded, Multiple Dose, Parallel Arm, Phase I Pilot Study of OXP001 Ibuprofen 400 mg Tablets and Brufen 400 mg Tablets in Normal, Healthy, Adult, Human Subjects Under Fasting Conditions to Assess The Incidence of Upper Gastrointestinal Irritation
Brief Title: Pilot Study of OXP001 and Brufen in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oxford Pharmascience Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OXP001-002
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: NSAID Related Gastric Irritation
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OXP001 (Experimental): OXP001
  Interventions: Drug: OXP001
- Ibuprofen (Active Comparator): Brufen
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: OXP001
  Arms: OXP001
Drug: Ibuprofen
  Other Names: Brufen
  Arms: Ibuprofen

SUMMARY:
Oxford Pharmascience (the sponsor) is developing a new formulation of Ibuprofen (OXP001 - the study drug) which it is proposed will have less of the side effects than are currently reported with standard prescription strength Ibuprofen.

This study will compare the study drug to an already marketed formulation of prescription strength Ibuprofen (the reference product) by looking at how the drug is taken up by the body and also by performing a specialist procedure called an endoscopy (or more specifically a gastroscopy). The safety and tolerability of the study drug will also be assessed.

The study will involve approximately 44 healthy male and female subjects. Subjects will be randomly assigned to receive either the study drug or reference product for 8 days. On Day 1, subjects will receive a single 800 mg dose of ibuprofen. On Days 2 to 9, subjects will receive 800 mg ibuprofen three times a day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Aged 18-55 years
* Normal, healthy upper gastrointestinal tract

Exclusion Criteria:

* History of or concurrent gastric irritation or ulcers
* History of allergy to non-steroidal anti-inflammatory drugs (NSAIDs)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2014-02; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Gastric irritation as measured by a Lanza score | 7 days

SECONDARY OUTCOMES:
Number of erosions | 7 days
Number of ulcers | 7 days
Incidence of gastric irritation | 7 days
Lanza score in stomach and duodenum | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mair, MB ChB, Principal Investigator — Quotient Clinical Ltd
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom